CLINICAL TRIAL: NCT02122926
Title: Effects of an Intensive Discharge Intervention on Medication Adherence, Glycemic Control, and Readmission Rates in Patients With Type 2 Diabetes
Brief Title: Intensive Discharge Intervention in Diabetes
Acronym: IDID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Jeffrey L. Schnipper, MD.,MPH., Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2010A056508; 2011-P-000217 (Other: Partners Human Research Committee)
Record Dates: First submitted 2013-01-25; First posted 2014-04-25 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Type II Diabetes; Cardiovascular Disease
Keywords: Transitions in care; discharge intervention; RCT; readmission rates; medication adherence; glycemic control; ED visits; medication reconciliation; Coleman Transitions Coach; telemonitoring; hypoglycemic events
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Medication Adherence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive discharge intervention (Experimental): The intervention is a multi-modal program consisting of the following:
  1. Inpatient protocol for adjusting the discharge diabetes regimen;
  2. Nurse practitioner "discharge advocate" to schedule follow-up appointments, prepare an after-hospital care plan, and patient education and counseling;
  3. Inpatient pharmacist counseling (identifying and addressing previous barriers to medication adherence, performing enhanced medication reconciliation, and patient education);
  4. Visiting nurse intervention after discharge;
  5. Follow-up in a post-discharge clinic with the NP discharge advocate and pharmacist /certified diabetes educator within 3 days of discharge;
  6. Telemonitoring of POC glucose levels to the study CDE, patient's PCP, or endocrinologist as appropriate; and
  7. Follow-up with PCP or endocrinologist within 1 week of discharge.
  Interventions: Other: Intensive discharge intervention
- Usual Care (No Intervention): Patients in the control arm of this study receive usual care.

INTERVENTIONS:
Other: Intensive discharge intervention — The intervention is a multi-modal program consisting of the following:
  1. Inpatient protocol for adjusting the discharge diabetes regimen;
  2. Nurse practitioner "discharge advocate" to schedule follow-up appointments, prepare an after-hospital care plan, and patient education and counseling;
  3. Inpatient pharmacist counseling (identifying and addressing previous barriers to medication adherence, performing enhanced medication reconciliation, and patient education);
  4. Visiting nurse intervention after discharge;
  5. Follow-up in a post-discharge clinic with the NP discharge advocate and pharmacist /certified diabetes educator within 3 days of discharge;
  6. Telemonitoring of POC glucose levels to the study CDE, patient's PCP, or endocrinologist as appropriate; and
  7. Follow-up with PCP or endocrinologist within 1 week of discharge.
  Arms: Intensive discharge intervention

SUMMARY:
The goal of this study is to design and implement an intensive discharge intervention for inpatients with type 2 diabetes and cardiovascular disease, and determine the effects of the intervention on post-discharge insulin adherence, glycemic control, cardiac medication adherence, hypoglycemic events, and emergency department visits and hospital readmissions.

ELIGIBILITY:
Inclusion Criteria:

* Adult inpatients at BWH on the medicine or cardiology services with a primary care physician who belongs to a participating practice or has not explicitly opted out of the study
* Type 2 diabetes
* Active cardiovascular disease
* Likely to be discharged home, and one of the following:

  1. prescribed insulin prior to admission
  2. prescribed two oral agents and with an A1c > 8.0 within 30 days of admission. - Practices that have already agreed to participate in this study for all their eligible patients.

Exclusion Criteria:

1. Discharge to a location other than home or rehabilitation (or to a caregiver's home)
2. Patient does not administer own medications and absence of a caregiver who lives with patient and administers all medications
3. Police custody, no telephone or homeless
4. Previous enrolment in the study within 90 days of discharge
5. Patient unable to communicate in either English or Spanish
6. Participation in the Integrated Care Management Program (iCMP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-12; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Cardiac medication adherence | 30 days after discharge
  Cardiac medication adherence as determined by patient self report 30 days after discharge

SECONDARY OUTCOMES:
Glycemic control | 90 days after discharge
  Glycemic control as determined by change in A1c 90 days after discharge.
Emergency department visits | Within 30 days after discharge
  Emergency department visits within 30 days of discharge.
Number of self-reported hypoglycemic events | Within 30 days of discharge
  Number of self-reported hypoglycemic events within 30 days of discharge.
Number of patient-days with hypoglycemia | Within 30 days of discharge
  Number of patient-days with hypoglycemia (point-of-care glucose less than 70 mg/dL) or with severe hypoglycemia (less than 40 mg/dL) within 30 days of discharge
Cardiac medication adherence | 90 days after discharge
  Cardiac medication adherence as determined by pharmacy refill rates for 90 days after discharge.
Hospital Readmissions | Within 30 days of discharge
  Hospital readmissions within 30 days of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Schnipper, MD, MPH, FHM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States